CLINICAL TRIAL: NCT06337214
Title: A Holistic Medical Approach - The Effect of "Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy" on Breast Cancer Patients Undergoing Cancer Therapy
Brief Title: TCM Therapy Program Impact on Breast Cancer Patients' Vital Energy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Attending physician of the hospital, Taipei City Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: TCHIRB-11301014-E
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Neoplasm, Breast; Patient Participation; Mental Health Issue
Keywords: Breast Cancer; Reinforcing Vital Energy; Patients Association; Patients Educatioin
MeSH Terms: conditions — Breast Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy (Experimental): This study aims to evaluate whether the participation in Traditional Chinese Medicine (TCM) supportive therapy courses, specifically the "Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy" , can enhance the quality of life of breast cancer patients undergoing treatment, increase their understanding and satisfaction with TCM adjunctive treatments, and bolster their confidence in cancer recovery. Evaluations will be conducted using pre- and post-tests spaced 4 to 6 weeks apart, during which participants will be administered three questionnaires.
  Interventions: Behavioral: Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy

INTERVENTIONS:
Behavioral: Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy — Comparing cancer patients who have participated in the program with those who have not, this study will examine differences in two types of quality of life questionnaires and constitution between the two groups.

SUMMARY:
The goal of this study is to evaluate the impact of the "Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy" on patients with breast cancer who are currently undergoing conventional Western medical treatments in Taiwan. The main questions it aims to answer are:

Can the "Traditional Chinese Medicine Therapy Program" alleviate symptoms experienced by breast cancer patients? Does the program improve the quality of life for breast cancer patients receiving Western medical treatments? How does the program contribute to the management of side effects associated with Western oncological therapies?

Participants will:

Engage in the "Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy" provided by the Taiwan Compassionate Cancer Care Association.

Receive supportive and educational services, including auxiliary Chinese medicine treatment courses, lifestyle and health education, and psychological counseling.

This study seeks to integrate the concept of holistic healthcare, emphasizing coordinated care that encompasses physical, mental, and social aspects, into the treatment of breast cancer.

DETAILED DESCRIPTION:
This study aims to evaluate whether the participation in Traditional Chinese Medicine (TCM) supportive therapy courses, specifically the "Traditional Chinese Medicine Therapy Program for Reinforcing Vital Energy" combined with the use of the herbal formulation at Taipei City Hospital, can enhance the quality of life of breast cancer patients undergoing treatment, increase their understanding and satisfaction with TCM adjunctive treatments, and bolster their confidence in cancer recovery.

This study adopts a holistic healthcare approach, integrating the Traditional Chinese Medicine (TCM) formulation Kuan-Sin-Yin from Taipei City Hospital with the "TCM Therapy Program for Reinforcing Vital Energy" course offered by a cancer patient support organization, to research its effects on breast cancer patients undergoing conventional medical treatment. International standard questionnaires and other inquiries are utilized to evaluate the impact on patients' physical, emotional, spiritual, and social well-being.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and above and below 85 years, willing to voluntarily participate in the study.
* Diagnosed with malignant breast tumors, ICD-10: C50, by conventional medicine.
* Patients currently undergoing cancer treatment, including chemotherapy, radiotherapy, or targeted therapy.

Exclusion Criteria:

* Diagnosed solely with carcinoma in situ or benign tumors, including fibrocystic breast conditions, by conventional medicine.
* Patients regularly receiving Astragalus polysaccharide injections.
* Patients with a history of allergies to Traditional Chinese Medicine.
* Pregnant or breastfeeding women.
* Individuals with a drug addiction habit, including both narcotic and non-narcotic drugs.
* Any other situation where the participant is unable to cooperate (e.g., due to any factor that prevents participation, deemed unsuitable for participation by study staff, unwillingness to sign the consent form).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire: Constitution in Chinese Medicine Questionnaire | Pre-test → Participation in "Traditional Chinese Medicine Program for Reinforcing Vital Energy" or not → Post-test After 4 ~6 weeks
  Observation and analysis Traditional Chinese Medicine Constitutions in breast cancer undergoing treatment
Questionnaire: Functional Assessment of Cancer Therapy-General Scale, FACT-G)(Version 4) | Pre-test → Participation in "Traditional Chinese Medicine Program for Reinforcing Vital Energy" or not → Post-test After 4 ~6 weeks
  Observation and analysis to measure four domains of QoL in cancer patients: Physical, social, emotional, and functional well-being
Questionnaire: European Organisation for Research and Treatment of Cancer, EORTC QLQ-BR23) | Pre-test → Participation in "Traditional Chinese Medicine Program for Reinforcing Vital Energy" or not → Post-test After 4 ~6 weeks
  Observation and analysis for measuring the quality of life in patients with breast cancer

SECONDARY OUTCOMES:
Additional questions regarding the "Traditional Chinese Medicine Program for Reinforcing Vital Energy" | Pre-test → Participation in "Traditional Chinese Medicine Program for Reinforcing Vital Energy" or not → Post-test After 4 ~6 weeks
  Understanding and Course satisfaction and Confidence in cancer recovery

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD. PhD, Study Director — Linsen, Chinese Medicine and Kunming Branch, Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan